CLINICAL TRIAL: NCT03592433
Title: Supporting Cancer Survivors' Health Insurance Marketplace Decisions
Brief Title: Improving Cancer Patients' Insurance Choices
Acronym: I Can PIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 201704045
Record Dates: First submitted 2018-06-26; First posted 2018-07-19 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Cancer; Health Literacy; Health Insurance; Health Services Accessibility; Informed Decision Making
Keywords: Decision Making; Decision Support; Health Literacy
MeSH Terms: conditions — Neoplasms | interventions — Decision Support Techniques

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- I Can PIC (Experimental): The I Can PIC website will be provided to participants randomized to the experimental/intervention group.
  Interventions: Behavioral: I Can PIC
- Attention Control (No Intervention): Participants randomized to the attention control group will be provided a link to a website developed by the American Cancer Society Cancer Action Network.

INTERVENTIONS:
Behavioral: I Can PIC — Participants will be shown (on a computer or via email link) a website called I Can PIC. I Can PIC provides health insurance education, suggests ways to learn about the costs of cancer care and follow-up, shows resources to help offset the high costs of care, and helps individuals estimate (based on national data) how much they might spend on health insurance in the upcoming year.
  Other Names: Decision Aid (DA)
  Arms: I Can PIC

SUMMARY:
The goal of this research study is to find out if a decision aid (DA) created by investigators, I Can PIC, is effective in helping cancer patients make decisions about their health insurance. The investigators will evaluate I Can PIC compared to an attention control condition (existing website created by the American Cancer Society Cancer Action Network). The study hypothesis is that those randomly assigned to I Can PIC will have higher knowledge about health insurance terms and details, more certainty about the best health insurance plan for them, and more confidence in their health insurance decisions compared to those randomly assigned to the control condition.

DETAILED DESCRIPTION:
In a prior study, the investigators created a consumer-friendly online tool, Show Me Health Plans (SMHP), for those enrolling in health insurance in the ACA marketplace. I Can PIC was developed based on SMHP, with input from an advisory board, and incorporating feedback from semi-structured qualitative interviews with cancer survivors. The investigators created I Can PIC to focus on unique needs of cancer patients and survivors considering health insurance. In this study, the investigators will examine the effectiveness of I Can PIC by conducting a randomized experiment with 275 participants. The trial will compare the I Can PIC to an attention control website developed by the American Cancer Society Cancer Action Network. Primary outcomes include knowledge, decision self-efficacy, certainty about plan choice, and the match between plan choice and preferences. The investigators will also explore whether financial toxicity, cancer type, and time since diagnosis relate to outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Ability to read English
* Diagnosed with cancer in the past 5 years
* Residing in Missouri or Illinois

Exclusion Criteria:

* Eligible for Medicaid or Medicare in Missouri or Illinois
* Enrolled in the following types of health insurance plans: Medicare, Medicaid, TRICARE or other military healthcare, or Indian Health Services

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 263 (Actual)
Dates: Start 2018-06-27 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Knowledge Score | Completed immediately after using I Can PIC
  The percent correct out of eight questions that were created by the research team based on information that is considered vital to making health insurance decisions.
Decision Self-efficacy | Completed immediately after using I Can PIC.
  The validated decision self-efficacy scale will be used. This 11-item scale measures an individual's self-confidence or belief in their ability to make a decision. Individuals will be asked to rate how confident they feel taking actions involved in making an informed choice (e.g., gathering information, asking questions, and expressing opinions).
Certainty about Choice (Decisional Conflict Scale) | Completed immediately after using I Can PIC
  The validated, 4-item SURE Test for clinical practice will be used. This scale measures whether individuals feel they have enough information to make a choice, are clear about their values for risks and benefits of their choice, and feel they have enough support to make a choice.

SECONDARY OUTCOMES:
Health Insurance Literacy Measure | Completed immediately after using I Can PIC
  Two items from the validated Health Insurance Literacy Measure will be used. This scale measures consumers' confidence in their ability to estimate their annual health care costs and their understanding of health insurance terms.
Health Insurance Literacy Measure | 3 month follow-up
  Two items from the validated Health Insurance Literacy Measure will be used. This scale measures consumers' confidence in their ability to estimate their annual health care costs and their understanding of health insurance terms.
  This measure will be assessed at follow-up to see if differences observed between groups immediately post-intervention, remain at follow-up.
Choice of Health Insurance Plan | Completed immediately after using I Can PIC
  Participants will be asked what health insurance plan they would choose. Plan selections will be categorized by the type of plan, e.g., high deductible plan, PPO, silver-tier Marketplace plan, gold-tier Marketplace plan, and will be compared to our algorithmic prediction about good fit plans for users based on estimates of their health care expenses.
Choice of Health Insurance Plan | 3 month follow-up
  Participants will be asked what health insurance plan they choose. Plan selections will be categorized by the type of plan, e.g., high deductible plan, PPO, silver-tier Marketplace plan, gold-tier Marketplace plan, and will be compared to our algorithmic prediction about good fit plans for users based on estimates of their health care expenses.
  This measure will be assessed at follow-up to see if differences observed between groups immediately post-intervention, remain at follow-up.
Healthcare Utlization | 3 month follow-up
  Participants will be asked questions about how often they use healthcare services to see if their plan choice relates to their utilization
Knowledge Score | 3 month follow-up
  The percent correct out of eight questions that were created by the research team based on information that is considered vital to making health insurance decisions.
  This measure will be assessed at follow-up to see if differences observed between groups immediately post-intervention, remain at follow-up.
Certainty about Choice (Decisional Conflict Scale) | 3 month follow-up
  The validated, 4-item SURE Test for clinical practice will be used. This scale measures whether individuals feel they have enough information to make a choice, are clear about their values for risks and benefits of their choice, and feel they have enough support to make a choice.
  This measure will be assessed at follow-up to see if differences observed between groups immediately post-intervention, remain at follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Mary C Politi, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Housten AJ, Furtado K, Kaphingst KA, Kebodeaux C, McBride T, Cusanno B, Politi MC. Stakeholders' perceptions of ways to support decisions about health insurance marketplace enrollment: a qualitative study. BMC Health Serv Res. 2016 Nov 8;16(1):634. doi: 10.1186/s12913-016-1890-8. PMID 27821121
- [Background] Politi MC, Barker AR, Kaphingst KA, McBride T, Shacham E, Kebodeaux CS. Show Me My Health Plans: a study protocol of a randomized trial testing a decision support tool for the federal health insurance marketplace in Missouri. BMC Health Serv Res. 2016 Feb 16;16:55. doi: 10.1186/s12913-016-1314-9. PMID 26880251
- [Background] Politi MC, Kuzemchak MD, Liu J, Barker AR, Peters E, Ubel PA, Kaphingst KA, McBride T, Kreuter MW, Shacham E, Philpott SE. Show Me My Health Plans: Using a Decision Aid to Improve Decisions in the Federal Health Insurance Marketplace. MDM Policy Pract. 2016 Jul;1(1):2381468316679998. doi: 10.1177/2381468316679998. Epub 2016 Nov 16. PMID 28804780
- See also: Decisional Conflict Scale Measure — https://decisionaid.ohri.ca/eval_dcs.html
- See also: Decision Self-Efficacy Scale Measure — https://decisionaid.ohri.ca/docs/develop/User_Manuals/UM_Decision_SelfEfficacy.pdf
- See also: Health Insurance Literacy Measure (HILM) — https://aircpce.org/projects/publications/development-health-insurance-literacy-measure-hilm-conceptualizing-and
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu